CLINICAL TRIAL: NCT03075605
Title: PROOF: Pancreatitis-associated Risk Of Organ Failure
Acronym: PROOF
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, David Whitcomb, Professor of Medicine, University of Pittsburgh
Other Study IDs: PRO08010374
Record Dates: First submitted 2017-02-02; First posted 2017-03-09 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Pancreatitis; Organ Failure, Multiple
MeSH Terms: conditions — Pancreatitis; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and DNA and urine samples will be collected and stored without personal identifiers (e.g. using a unique laboratory number or bar code) for future research involving pancreatic diseases to include pancreatitis and pancreatic cancer. Stored biospecimens collected for htis protocol may be shared in a de-identified manner with outside investigators with the approval of the principal investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Subjects with acute pancreatitis: Subjects with acute pancreatitis
- Subjects with previous attack: Subjects with previous attack
- Controls: Controls

SUMMARY:
This is a prospective case control study that compares the initial immune response with severity and outcome in patients with acute pancreatitis.

DETAILED DESCRIPTION:
This is a prospective case control study that compares the initial immune response with severity and outcome in patients with acute pancreatitis. Therefore, the investigators aim to determine whether etiology of acute pancreatitis, segregates with candidate genetic polymorphisms and their m-RNA expression, as well as whether functional polymorphisms in inflammation regulating genes predict a more severe outcome in acute pancreatits. The investigators anticipate that based on our results that we will provide a more accurate predictor of the clinical course of acute pancreatits and help direct more aggressive or cytokine specific treatment of patients at greater risk of a more severe form of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for Subjects (all three) Males and females of 16 years of age and older. Body weight at least 40kg

Diagnosis of acute pancreatitis by both: Abdominal pain or abdominal localizing signs AND Elevated amylase levels by at-least three times the upper limit of normal and/or elevated lipase levels by at-least three times the upper limit of normal (25, 26). Acute pancreatitis must be defined by 2 of the 3 following criteria:

* Serum amylase or lipase elevated greater than 3X upper limit of normal
* epigastric acute pancreatitis pain
* abdominal imaging studies demonstrating pancreatic edema, peripancreatic fat stranding or complications or acute pancreatitis Willingness to participate in the study and sign the informed consent. (Children and subjects who are cognitively impaired for temporary reasons as mentioned in the section 4.7 of this protocol will require a representative to sign the informed consent).

Inclusion criteria for Controls (all three) Males and females of 18 years of age and older. a. Unrelated family member or a friend of the subject or a patient having blood drawn in general medicine outpatient clinic, without a history of pancreatitis, OR Willingness to participate in the study and sign the informed consent.

Additional Inclusion Criteria for subjects with a previous attack of acute pancreatitis:

age criteria as defined above.

- Previous severe attack of severe acute pancreatitis requiring a ICU stay of at least 48 hours or evidence of pancreatic necrosis on computerized tomography.

Willingness to participate and sign informed consent

Exclusion Criteria:

* Exclusion Criteria for Subjects:

Persons unwilling to sign the informed consent Disorientation secondary to irreversible organic brain damage. Mean corpuscular volume (MCV) of less than 77 in all children of 18 years or younger.

Blood transfusion within one week of enrollment Chronic Pancreatitis History of pancreatic cancer History of cancer requiring chemotherapy or radiation within the past 1 year History of organ transplant Subject is a prisoner Pancreatitis due to multiple trauma or surgical complications

Exclusion criteria for Controls:

Persons unwilling to sign the informed consent

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Both males and females, over 1 year of age.
Sampling Method: Probability Sample
Enrollment: 723 (Actual)
Dates: Start 2008-05-20 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Severe Acute Pancreatitis (defined as persistent organ failure) | 1 year
  To compare the initial immune response in patients who developed mild vs. severe disease. To determine whether functional polymorphisms in inflammation regulating genes predicts a more severe outcome in acute pancreatitis.

CONTACTS AND LOCATIONS:
Overall Officials: George Papachristou, MD, Study Chair — Ohio State University

IPD SHARING:
Plan to Share IPD: Undecided
If shared, all individual identifiers will be removed.

REFERENCES:
- [Derived] Langmead C, Lee PJ, Paragomi P, Greer P, Stello K, Hart PA, Whitcomb DC, Papachristou GI. A Novel 5-Cytokine Panel Outperforms Conventional Predictive Markers of Persistent Organ Failure in Acute Pancreatitis. Clin Transl Gastroenterol. 2021 May 6;12(5):e00351. doi: 10.14309/ctg.0000000000000351. PMID 33955376
- [Derived] Komara NL, Paragomi P, Greer PJ, Wilson AS, Breze C, Papachristou GI, Whitcomb DC. Severe acute pancreatitis: capillary permeability model linking systemic inflammation to multiorgan failure. Am J Physiol Gastrointest Liver Physiol. 2020 Nov 1;319(5):G573-G583. doi: 10.1152/ajpgi.00285.2020. Epub 2020 Sep 2. PMID 32877220
- [Derived] Dugum M, Gougol A, Paragomi P, Gao X, Matta B, Yazici C, Tang G, Greer P, Pothoulakis I, O'Keefe SJD, Whitcomb DC, Yadav D, Papachristou GI. Association of Dietary Habits with Severity of Acute Pancreatitis. Curr Dev Nutr. 2018 Oct 8;2(12):nzy075. doi: 10.1093/cdn/nzy075. eCollection 2018 Dec. PMID 30569031